CLINICAL TRIAL: NCT01291355
Title: Maternal Positioning to Correct Occipitoposterior Fetal Position in Labor: A Randomized Controlled Trial
Brief Title: Maternal Positioning and Occipitoposterior Fetal Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Applied Sciences of Western Switzerland (Other); Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Marie-Julia GUITTIER, RM, PhD, University of Applied Sciences of Western Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER10-042
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Maternal Distress in Labor; Persistent Occipitoposterior or Occipitoanterior Position; Dystocia; Fetal Position and Presentation Abnormalities
Keywords: Maternal position; Occipitoposterior position; Labor; Dystocia; Fetal presentation Abnormalities
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Specific maternal position (Experimental): women allocated to intervention group will be invited to adopt a posture all fours type:"support on the knees, torso tilted forward, back stretched" for a minimum of 10 minutes. A cushion is placed between the legs of the woman to limit the cuts. According to Dr de Gasquet, author of the description of this posture, the effect on the variety of presentation would be almost immediate.
  Interventions: Other: Specific maternal position during the labor
- Control (No Intervention): Not specific intervention for this group- Only usual care

INTERVENTIONS:
Other: Specific maternal position during the labor — women allocated to intervention group will be invited to adopt a posture all fours type:"support on the knees, torso tilted forward, back stretched" for a minimum of 10 minutes. A cushion is placed between the legs of the woman to limit the cuts.
  Arms: Specific maternal position

SUMMARY:
The aim of the study is to evaluate the efficacy of a specific maternal position to correct fetal position in occipito-posterior during the labor.

The investigators hypothesize that the maternal position described by the Dr de Gasquet facilitate the rotation in occipito-anterior during the labor.

The calculated sample size is 438 participants (219 in each group)

DETAILED DESCRIPTION:
Randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* singleton
* primiparous and multiparous
* Term ≥ 37 weeks
* Labor in dilatation phase (cervix effaced, permeable finger 2 to 9 cm)
* Diagnosis of occipitoposterior variety confirmed by ultrasound

Exclusion Criteria:

* Maternal age below 18 years old
* Misunderstanding the French Language
* Full dilatation of the cervix
* Posture evaluated already adopted by the woman during labor

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 438 (Actual)
Dates: Start 2011-02; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Fetal presentation after the intervention compare to control group | One hour after the randomization for the study
  Diagnosis of the fetal presentation will be measured by an ultra-sound one hour after the randomization in both groups: intervention and control

SECONDARY OUTCOMES:
Maternal comfort and pain sensation | During the hour after the randomization
  Auto-administrated questionnaire to assess comfort of the maternal position and pain related to the labor, in intervention group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Julia GUITTIER, PhD, Principal Investigator — University Hospitals of Geneva-Switzerland
Locations (2):
- Switzerland (2):
  - Maternity of University Hospitals, Geneva
  - University Hospitals - Maternity, Geneva

REFERENCES:
- [Result] Guittier MJ, Othenin-Girard V, Irion O, Boulvain M. Maternal positioning to correct occipito-posterior fetal position in labour: a randomised controlled trial. BMC Pregnancy Childbirth. 2014 Feb 24;14:83. doi: 10.1186/1471-2393-14-83. PMID 24564746
- [Result] Guittier MJ, Othenin-Girard V. [Correcting occiput posterior position during labor: the role of maternal positions]. Gynecol Obstet Fertil. 2012 Apr;40(4):255-60. doi: 10.1016/j.gyobfe.2011.05.006. Epub 2011 Nov 17. French. PMID 22099975